CLINICAL TRIAL: NCT05522205
Title: WEED CARE - Randomized Controlled Study on Regulated Cannabis Access for Recreational Use in Pharmacies in Basel
Brief Title: Regulated Cannabis Access in Basel
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health Department of the Canton of Basel-Stadt (Other Government)
Collaborators: University of Basel (Other); University Psychiatric Clinics Basel (Network); Psychiatric Services Aargau AG (Other)
Responsible Party: Principal Investigator, Marc Walter, Prof. Dr. med., Psychiatric Services Aargau AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-01670
Record Dates: First submitted 2022-08-08; First posted 2022-08-30 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Cannabis Use Disorder; Mental Health Disorder; Physical Illness
Keywords: cannabis regulation; health effects; cannabis consumption
MeSH Terms: conditions — Mental Disorders | interventions — Pharmacies

STUDY DESIGN:
Masking Description: One group has immediately access to regulated cannabis access in pharmacies and the other group has to wait six months until they have regulated cannabis access.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Immediately regulated cannabis access in pharmacies.
  Interventions: Other: Regulated cannabis access in pharmacies
- Control group (No Intervention): During the first six months participants of the control group have to continue to buy their cannabis on the illicit market. Afterthese six months they also have access to regulated cannabis access.

INTERVENTIONS:
Other: Regulated cannabis access in pharmacies — The study does not investigate the health effects of cannabis. The study investigates the effects of regulated cannabis access on cannabis consumption and health in comparison to the unregulated illegal market.
  Arms: Experimental group

SUMMARY:
The randomised controlled study on regulated cannabis access in pharmacies in Basel aims to investigate the effects of regulated cannabis access on consumption behaviour and mental and physical health in comparison to the illegal market.

DETAILED DESCRIPTION:
This project consist of two parts: The first part is a randomised controlled study, the second part is an observational study. The randomised controlled study will last six months. Participants will randomly be assigned to one of two groups: Group 1 has immediately access to regulated cannabis in pharmacies; Group 2 has to wait for six months. After six months all participants will have access to regulated cannabis in pharmacies (oberservational study). Every six month participants will be invited to answer online-questionnaires on their cannabis consumption behavior, their mental and physical health. The entire study lasts 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years, residence in Basel-Stadt, consuming cannabis at least monthly during the last 6 months (positive urine sample)

Exclusion Criteria:

* pregnant or breastfeeding, currently suicidal, currently psychotic, current inpatient psychiatric treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in problematic cannabis consumption behaviour | 6 / 12 /18 /24 / 30 months
  Cannabis Use Disorder Identification Test - Revised; min. value 0, max. value 32; higher scores mean worse outcome

SECONDARY OUTCOMES:
Change in depression | 6 / 12 /18 /24 / 30 months
  Patient Health Questionnaire; min. value 0, max. value 27; higher scores mean worse outcome
Change in anxiety | 6 / 12 /18 /24 / 30months
  Generalized Anxiety Disorder; min. value 0, max. value 21; higher scores mean worse outcome
Change in psychosis | 6 / 12 /18 /24 / 30 months
  Checklist of early intervention; min. value 0, max. value 8; higher scores mean worse outcome
Change in physical health | 6 / 12 /18 /24 / 30 months
  Symptom Checklist - 90, Somatization; min. value 0, max. value 48; higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Canton Basel-Stadt, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publications.
Supporting Information: SAP, ICF
Time Frame: 6 months after publication
Access Criteria: Only research institutions will have access. Data dictionaries will be shared for studies that are planning to investigate similar research questions. Principal investigator or co-investigator will review the requests.

REFERENCES:
- [Derived] Baltes-Flueckiger L, Steinauer R, Meyer M, Vogel M, Walter M. Effects of cannabis regulation in Switzerland: Study protocol of a randomized controlled trial. Front Psychiatry. 2023 Mar 23;14:1139325. doi: 10.3389/fpsyt.2023.1139325. eCollection 2023. PMID 37032954